CLINICAL TRIAL: NCT02495961
Title: Study of Chronic Degenerative Diseases, Translational Medicine Approach
Brief Title: Study of Chronic Degenerative Diseases
Status: Completed | Type: Observational
Sponsor: Asociación Científica Latina A.C. (Other)
Collaborators: Universidad Autonoma del Estado de Mexico (Other); Ciprés Grupo Médico CGM SC (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-01
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Metabolic Syndrome X
Keywords: hyperlipidemias; hyperglycemia; hypertension; leptin; hyperhomocysteinemia
MeSH Terms: conditions — Metabolic Syndrome; Hyperlipidemias; Hyperglycemia; Hypertension; Hyperhomocysteinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low risk population: Colombian children, between 6 and 12 years old, regular students of a Primary school.
- High risk population: Mexican children, between 6 and 12 years old, regular students of a Primary school.

SUMMARY:
The prevalence of obesity and type 2 diabetes mellitus (DM) in children have been increasing in parallel at an alarming rate. In particular, the increasing prevalence of type 2 DM is attributable to genetic factors, clinical (waist circumference, adiposity and physical condition) and biochemical (insulin secretion and sensitivity, lipids and inflammation) risk, each of which represents an independent risk.

As has already studied and published in the investigators' group, the child population of Toluca has greater expression of cardiovascular risk factors than their counterparts in Bogota, Colombia. The metabolic characterization of the young population of Toluca and Bogota with new biomarkers such as homocysteine and leptin is an activity that aims to provide more metabolic data affecting young people.

Hypothesis:

After six months of follow-up there will be a greater relative risk in Mexican population to have identified another component of metabolic syndrome compared to the young population of Colombia.

DETAILED DESCRIPTION:
Objective:

To compare the expression levels of cardiovascular risk markers in young people between 5 and 12 years of Toluca, Mexico and Bogota, Colombia.

Material and methods:

Type of study: prospective, descriptive, comparative, and longitudinal.

Sample Calculation:

For a cohort study and taking into account that in the investigators' previous publication in the Colombian population only 13% (sick rate in unexposed group) had an altered metabolic parameter; accepting an alpha risk of 0.05 and a beta of 0.2 on a risk bilateral contrast, 57 subjects were required in the exposed group (Mexican population) and 57 in unexposed to detect a minimum relative risk of 3 to find other alteration to metabolic syndrome after six months follow-up.

Measurements:

The International Physical Activity Questionnaire (IPAQ) will be applied to all children. Dietary history of three days and physical examination (height in cm , weight in kg and waist circumference in centimeters) and blood pressure (mmHg) data will be recorded. Blood samples will be taken to analyze glucose, cholesterol, HDL, triglycerides, homocysteine and leptin.

Statistics:

Variables will be tested for normality through the Kolmogorov-Smirnov and Shapiro-Wilk formulas. Variables related to the physiological and metabolic functions and anthropometric measurements will be reported in mean and standard deviation. The differences in the laboratorial and anthropometrical variables will be analyzed with the Student t test. A difference will be considered significant with a p value ≤ 0.05. The statistical program used is the Statistical Package for the Social Sciences (SPSS) version 19.

ELIGIBILITY:
Inclusion Criteria:

* Primary school students of medium-low income.

Exclusion Criteria:

* Children with disabilities or a known chronic disease.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary school students.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome component detection | six months
  After six months of a basal evaluation, children will be re-examined in each component of the metabolic syndrome.
  Metabolic syndrome component detection will be determined by the measure of glucose (mg/dl), cholesterol (mg/dl), triglycerides (mg/dl), high-density lipoproteins (HDL), waist circumference (cm), hip circumference (cm) and blood pressure (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD., Principal Investigator — Asociación Científica Latina A.C.
Locations (1):
- Asociación Científica Latina A.C., Toluca, State of Mexico, Mexico